CLINICAL TRIAL: NCT00363025
Title: A Randomized Multicenter Study of More Intensive Versus Less Intensive Post-Remission Therapy in Elderly Patients With Acute Myelogenous Leukemia (AML) or Transformed Refractory Anemia With Excess Blasts (RAEB-t).
Brief Title: A Randomized Study of Post-Remission Therapy in Elderly Patients With Acute Myelogenous Leukemia.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Acute Leukemia French Association (Other)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALFA-9803
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2006-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute myeloid leukemia; Older patients; Patient aged 65 years or more
MeSH Terms: conditions — Leukemia, Myeloid, Acute

INTERVENTIONS:
Procedure: Two post-remission strategies
Drug: Idarubicin versus daunorubicin

SUMMARY:
In this ALFA-9803 trial in AML patients aged 65 years or more, we randomly compared idarubicin or daunorubicin throughout the study (first randomization) and two different post-remission strategies (second randomization): one single intensive consolidation course similar to induction versus six ambulatory cycles with one dose of idarubicin/daunorubicin (day 1) and 2x60 mg/m2/d cytarabine SC (day 1 to 5) delivered in out-patients on a monthly basis. Primary endpoint was 2-year overall survival (OS). Study hypotheses were equivalence for the idarubicin/daunorubicin comparison and a 15% difference in 2-year OS for the post-remission therapy comparison.

DETAILED DESCRIPTION:
Patients were randomized at baseline (first R1 randomization) to receive either daunorubicin (DNR) or idarubicin (IDA) as an anthracycline for induction and post-remission therapy. This first randomization was stratified on centers and AML type (de novo versus post-MDS AML). Induction chemotherapy consisted of a 4+7 course with either DNR at a daily dosage of 45 mg/m2 or IDA at a daily dosage of 9 mg/m2 for four days (day 1 to day 4) in combination with 200 mg/m2 cytarabine per day as a continuous IV infusion for seven days (day 1 to 7). Lenograstim granulocyte colony-stimulating factor (G-CSF) was administered in all patients from day 9 until myeloid recovery (3 consecutive days with PMN more than 1.0 G/L) by IV infusion and at a daily dosage of 263 microg/day for a maximum of 28 days. A blood and marrow aspiration smear examination was performed at day 21. A salvage course of chemotherapy may be offered to patients with persistent leukemia (defined below), but only if they did not present acquired contra-indication to further intensive chemotherapy (baseline criteria). Salvage consisted of six 1-hour IV bolus of intermediate-dose cytarabine (500 mg/m2/12h day 1 to 3) combined to mitoxantrone (MTZ) at a daily dosage of 12 mg/m2 for two days (day 3 and 4). G-CSF administration was stopped before salvage onset and restarted from day 5 of the salvage course until myeloid recovery for a maximum of 28 days.

Patients reaching complete remission (CR) after induction or induction followed by salvage were eligible for a second R2 randomization between mild versus intensive post-remission therapy, but only if they did not present acquired contra-indication to further intensive chemotherapy (baseline criteria). This second randomization was stratified on centers, AML groups (de novo versus post-MDS AML), and first randomization groups. Mild post-remission therapy was administered in out-patients and consisted of six 1+5 monthly courses with either 45 mg/m2 DNR or 9 mg/m2 IDA for one day (day 1) in combination with 60 mg/m2/12h cytarabine as a SC infusion for five days (day 1 to 5). No G-CSF support was given after these six courses. Intensive post-remission therapy required another hospitalization and was a repetition of the first 4+7 induction administered at the same doses and followed by G-CSF administration as well.

ELIGIBILITY:
Inclusion Criteria:

Male or female aged 65 years or more. Patient with previously untreated AML except M3 in the FAB classification. Patient with previously untreated transformed refractory anemia with excess blasts (RAEB-t).

Patients with AML secondary to a previously untreated myelodysplastic syndrome (MDS), documented or not, are eligible, as well as those with RAEB-t evolving from a previous known MDS.

Patients with a Performance Status < 3. Patient who has given his/her written informed consent.

Exclusion Criteria:

Patients with AML3 in the FAB classification. Patients with blast crisis of previously known myeloproliferative syndrome. Patients with AML secondary to previous treatment with cytotoxic chemotherapy or radiotherapy (therapy-related AML).

Patients with another concommitant neoplasia. Patients with leukemic central nervous system involvement. Patients with a Grade > 2 uncontrolled infection. Patients with Grade > 2 visceral contra-indications to treatment with induction chemotherapy (except if leukemia-related).

Bilirubin > 2 times the normal range of the laboratory. Serum creatinine > 2 times the normal range of the laboratory. Patients with cardiac contra-indication to treatment with anthracyclines.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 465
Dates: Start 1999-11; Study Completion 2006-04

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Complete remission rate
Induction death rate

CONTACTS AND LOCATIONS:
Overall Officials: Herve Dombret, M.D., Principal Investigator — Acute Leukemia French Association
Locations (13):
- France (13):
  - Hopital Avicenne, Bobigny
  - Hopital Percy, Clamart
  - Hopital Henri Mondor, Créteil
  - CHU, Lille
  - CHU, Limoges
  - Hopital Edouard Herriot, Lyon
  - Hopital Pitie-Salpetriere, Paris
  - Hopital Saint-Louis, Paris
  - CHU, Rouen
  - CNLCC, Rouen
  - CNLCC, Saint-Cloud
  - CH, Versailles
  - IGR, Villejuif

REFERENCES:
- [Derived] Sarkozy C, Gardin C, Gachard N, Merabet F, Turlure P, Malfuson JV, Pautas C, Micol JB, Thomas X, Quesnel B, Celli-Lebras K, Preudhomme C, Terre C, Fenaux P, Chevret S, Castaigne S, Dombret H. Outcome of older patients with acute myeloid leukemia in first relapse. Am J Hematol. 2013 Sep;88(9):758-64. doi: 10.1002/ajh.23498. Epub 2013 Aug 7. PMID 23749683
- [Derived] Gardin C, Chevret S, Pautas C, Turlure P, Raffoux E, Thomas X, Quesnel B, de Revel T, de Botton S, Gachard N, Renneville A, Boissel N, Preudhomme C, Terre C, Fenaux P, Bordessoule D, Celli-Lebras K, Castaigne S, Dombret H. Superior long-term outcome with idarubicin compared with high-dose daunorubicin in patients with acute myeloid leukemia age 50 years and older. J Clin Oncol. 2013 Jan 20;31(3):321-7. doi: 10.1200/JCO.2011.40.3642. Epub 2012 Dec 17. PMID 23248249
- [Derived] Itzykson R, Gardin C, Pautas C, Thomas X, Turlure P, Raffoux E, Terre C, Fenaux P, Castaigne S, Dombret H, Boissel N; Acute Leukemia French Association (ALFA). Impact of post-remission therapy in patients aged 65-70 years with de novo acute myeloid leukemia: a comparison of two concomitant randomized ALFA trials with overlapping age inclusion criteria. Haematologica. 2011 Jun;96(6):837-44. doi: 10.3324/haematol.2010.036921. Epub 2011 Apr 1. PMID 21459791
- [Derived] Malfuson JV, Etienne A, Turlure P, de Revel T, Thomas X, Contentin N, Terre C, Rigaudeau S, Bordessoule D, Vey N, Gardin C, Dombret H; Acute Leukemia French Association (ALFA). Risk factors and decision criteria for intensive chemotherapy in older patients with acute myeloid leukemia. Haematologica. 2008 Dec;93(12):1806-13. doi: 10.3324/haematol.13309. Epub 2008 Oct 6. PMID 18838471